CLINICAL TRIAL: NCT04952324
Title: MTHFR Gene Mutation C6777T and Concentration of Vitamin B12, Folic Acid, Homocysteine and High Sensitive CRP in the Blood of Pregnant Women With Gestational Diabetes Mellitus.
Brief Title: MTHFR Mutation and Concentration of B12,Folic Acid,Homocysteine and HS CRP in the Blood of Pregnant Women With GDM.
Status: Completed | Type: Observational
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Ana Bošković, mr. sc. Ana Boskovic, Ob/Gyn specialist, University of Mostar
Other Study IDs: MTHFR mutation and GDM
Record Dates: First submitted 2021-05-31; First posted 2021-07-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection; Vitamin B 12; Folic Acid; C-Reactive Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Biospecimen Retention: Samples Without DNA — Periferal blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pregnant women with GDM: Pregnant women with GDM
  Interventions: Other: Blood sampling and determination of MTHFR mutation,vitamin B12, folic acid, homocystein and HS CRP
- Pregnant women without GDM: Pregnant women without GDM
  Interventions: Other: Blood sampling and determination of MTHFR mutation,vitamin B12, folic acid, homocystein and HS CRP

INTERVENTIONS:
Other: Blood sampling and determination of MTHFR mutation,vitamin B12, folic acid, homocystein and HS CRP — Periferal Blood sampling and determination of MTHFR mutation,vitamin B12, folic acid, homocystein and high sensitive CRP

SUMMARY:
Research hypothesis:

* pregnant women with gestational diabetes have elevated serum CRP values and homocysteine compared to pregnant women with normal glucose metabolism
* Elevated CRP and homocysteine values are associated with poorer perinatal outcome.
* reduced concentrations of folic acid and vitamin B 12 are associated with higher homocitein values
* Carriers of the MTHFR gene mutation have higher homocysteine concentrations

DETAILED DESCRIPTION:
Research issues:

The basic pathophysiological mechanism of gestational diabetes is insulin resistance formed as a result of the production of placental hormones. It turned out as atherosclerosis, chronic cardiovascular diseases and diabetes share common pathophysiological mechanisms, which is nonphysiological activation of the endothelium. CRP is an acute phase protein that is synthesized in the liver to stimulate IL-6. It is a sensitive marker of inflammation and good predictor of the development of preeclampsia while the research results CRP as a predictor of gestational diabetes inconsistent. Homocysteine is a marker of endothelial dysfunction and oxidative stress. Elevated homocysteine levels are a factor risk of cardiovascular disease, and in pregnancy is associated with preeclampsia, spontaneous abortions and placental abruption.Proper adjustment of uteroplacental blood vessels is necessary for the orderly course of pregnancy these deviations from normal endothelial function will lead to pregnancy disorders.

This study is an extrapolation of recognized markers of cardiovascular risk to gestational diabetes for the purpose of predicting an adverse perinatal outcome. Examined the association of the combination of the hs-CRP marker and homocysteine with gestational diabetes and pregnancy outcome and the correlation of homocysteine and folic acid concentration acid and vitamin B12.

Research hypothesis:

* pregnant women with gestational diabetes have elevated serum CRP values and homocysteine compared to pregnant women with normal glucose metabolism
* Elevated CRP and homocysteine values are associated with poorer perinatal outcome.
* reduced concentrations of folic acid and vitamin B 12 are associated with higher homocitein values
* Carriers of the MTHFR gene mutation have higher homocysteine concentrations

Research goals:

* compare serum values of hs-CRP and homocysteine in pregnant women with gestational diabetes and in the control group of pregnant women with a regular sugar load test
* determine the existence of an association between the values of hs-CRP and homocysteine with complications of pregnancy.
* determine the existence of a correlation between the values of vitamin B12 and folic acid with serum homocysteine values
* determine the association of MTHFR gene mutation and homocysteine concentration The objectives of the research are achievable by the proposed research.

Respondents:

* Study group: 100 pregnant women hospitalized for sugar profile in the Department pathology of pregnancy, Clinic for Gynecology and Obstetrics, SKB Mostar, and which was previously diagnosed with gestational diabetes
* Control group: 100 pregnant women with a regular glucose load test, and which meet the inclusion criteria

Criteria for inclusion in the research:

* Age of respondents from 18 to 35 years
* Single pregnancies BMI from 18.5 to 29.9 kg / m 2

Exclusion criteria:

* Diagnosis of acute and chronic inflammatory diseases
* Pregestational diabetes
* Chronic hypertension
* Multiple pregnancies
* Smoking

This enzyme is important for the metabolism of folate, B12, homocysteine.The diagnosis of gestational diabetes will be based on the results of the HAPO study, which is also accepted by the WHO. All respondents will be measured values of hs-CRP, homocysteine, folic acid and vitamin B12 in serum, at gestational age between 24-28 weeks of gestation and compare between test and control groups. The correlation of folate acid and vitamin B12 it will be examined the conection between homocysteine values in serum.

Using patients' medical histories we will monitore examined parameters: birth weight and length of the newborn, Apgar sum newborns in the 1st and 5th minutes, the development of hypertensive pregnancy disorders (hypertension, preeclampsia), HbA1c, BMI values and weight gain in pregnancy, gestational age, frequency of induced labor, cesarean section and surgically completed vaginal delivery, frequency of shoulder dystocia, presence meconium fruits, polyhydramnios, oligohydramnios and hypothyroidism. Statistical analysis of the data will assess the association of pregnancy outcomes with hs-CRP and homocysteine values in both study groups of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* age of respondents from 18 to 35 years
* Single pregnancies BMI from 18.5 to 29.9 kg / m 2

Exclusion Criteria:

* Diagnosis of acute and chronic inflammatory diseases
* Pregestational diabetes
* Chronic hypertension
* Multiple pregnancies
* Smoking

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Population of women who were hospitalized at the gynecology and obstretics clinic in Mostar.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Whether increased hs crp and homocysteine values are associated with poorer perinatal outcome | Between 24 and 28 weeks of gestation
  We will meassure hs CRP and homocysteine levels in pregnant women with GDM and compare to hs CRP and homocysteine levels in pregnant women with normal glucose metabolism
carriers of the MTHFR gene mutation have higher serum homocysteine concentrations in the blood | Between 24 and 28 weeks of gestation
  We will compare serum homocysteine levels in pregnant carriers of the MTHFR gene mutation and pregnant women normal MTHFR gene mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Vajdana Tomic, prof. dr, Study Chair — Faculty of Health Studies, Mostar
Locations (2):
- Bosnia and Herzegovina (2):
  - Faculty of health studies, Mostar, Mostar
  - University of Mostar, Mostar

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginnibg 3 months and ending 5 Years folowing article publication.
Access Criteria: Investigators whose proposed use the Data has been approved by an Independent review committee identified for this purpose.

REFERENCES:
- [Derived] Boskovic A, Cuk A, Mandrapa V, Dugandzic Simic A, Cvetkovic I, Orlovic Vlaho M, Kresic T, Tomic T, Tomic V. Association of MTHFR polymorphism, folic acid and vitamin B12 with serum homocysteine levels in pregnant women. Biomol Biomed. 2024 Jan 3;24(1):138-143. doi: 10.17305/bb.2023.9260. PMID 37622180
- See also: Chemical pathology of homocysteine. IV. Excitotoxicity, oxidative stress, endothelial dysfunction, and inflammation — https://pubmed.ncbi.nlm.nih.gov/19667406/
- See also: First-Trimester Screening for Gestational Diabetes Mellitus Based on Maternal Characteristics and History — https://pubmed.ncbi.nlm.nih.gov/25531073/
- See also: Endothelial dysfunction - a major mediator of diabetic vascular disease — https://pubmed.ncbi.nlm.nih.gov/23994612/
- See also: Inflammatory and Other Biomarkers: Role in Pathophysiology and Prediction of Gestational Diabetes Mellitus — https://pubmed.ncbi.nlm.nih.gov/26110385/